CLINICAL TRIAL: NCT03767751
Title: Phase I/II Study to Evaluate Treatment of Relapsed or Refractory Multiple Myeloma With Dual CAR-T Cells Targeting CD38 and BCMA
Brief Title: A Feasibility and Safety Study of Dual Specificity CD38 and BCMA CAR-T Cell Immunotherapy for Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Molecular & Immunological Department,Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-037
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Dual Specificity CD38 and bcma CAR-T Cells — 1) Biological: Dual Specificity CD38 and BCMA CAR-T Cells,2)1-5X10E6/Kg

SUMMARY:
CAR-T cell therapy has shown promising results for the treatment of relapsed or refractory Multiple Myeloma,however, a subset of patients relapse due to the loss of target in tumor cells.Dual Specificity CD38 and BCMA CAR-T cells can recognize and kill the malignant cells through recognition of CD38 or BCMA. This is a phase 1/2 study designed to determine the safety of dual specificity CD38 and BCMA CAR-T cells and the feasibility of making enough to treat patients with relapsed or refractory Multiple Myeloma.

DETAILED DESCRIPTION:
1. PRIMARY OBJECTIVES:

   1. To evaluate the feasibility and safety of dual specificity CD38 and BCMA CAR-T cells in patients with relapsed or refractory Multiple Myeloma.
   2. To evaluate the duration of in vivo persistence of adoptively transferred T cells, and the phenotype of persisting T cells.Real Time polymerase chain receptor (RT-PCR) and Flow cytometry(FCM) analysis of PB,BM and lymph node will be used to detect and quantify survival of universal dual specificity CD38 and BCMA CAR-T cells over time.
2. SECONDARY OBJECTIVES:

1.For patients with detectable disease, measure anti-tumor response due to dual specificity CD38 and BCMA CAR-T cell infusions.

2.The CAR-T cells will be administered by i.v. injection over 20-30 minutes as a using Day 0: 1-5x10e6/kg total dose on day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant
2. 12 Years to 70 Years (Child, Adult, Senior)
3. Patient with relapsed or refractory Multiple Myeloma,multiple myeloma cell express CD38(over 50%) and BCMA (over 50%)
4. Estimated life expectancy ≥ 12 weeks (according to investigator's judgement)
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
6. Adequate organ function

Exclusion Criteria:

1. Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease
2. Diagnosis of Burkitt's leukemia/lymphoma according to WHO classification or chronic myelogenous leukemia lymphoid blast crisis
3. Richter's syndrome
4. Presence of Grade II-IV (Glucksberg) or B-D (IBMTR) acute or extensive chronic GVHD at the time of screening
5. Subjects with any autoimmune disease or any immune deficiency disease or other disease in need of immunosuppressive therapy
6. Severe active infection (uncomplicated urinary tract infections, bacterial pharyngitis is allowed), Prophylactic antibiotic, antiviral and antifungal treatment is permissible
7. Active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening
8. Patient has an investigational medicinal product within the last 30 days prior to screening
9. Previous treatment with investigational gene or cell therapy medicine products
10. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
11. Pregnant or nursing women

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2022-12-05 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe/Adverse Events as a Measure of Safety and Tolerability | 24weeks
MTD of dual specificity CD38 and BCMA CAR-T cells | 4 weeks
  The highest dose of dual specificity CD38 and BCMA CAR-T cells that is estimated to result in defined Dose Limiting Toxicity (DLT) with the exception of allowable 'expected' AEs associated with the intravenous infusion of dual specificity CD38 and BCMA CAR-T cells
Copies numbers of CAR in peripheral blood(PB), bone marrow(BM)and lymph nodes | 24 weeks

SECONDARY OUTCOMES:
Six-month Objective response rate of complete remission and partial remission | 24 weeks
Six-month Overall survival | 24 weeks
Six-month Progression free survival | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Hematology Department of Chinese PLA General Hospital, Beijing, China